CLINICAL TRIAL: NCT03265769
Title: Femoral or Radial Approach in the Treatment of Coronary Chronic Total Occlusion: A Randomized Clinical Trial (FORT CTO TRIAL)
Brief Title: Femoral or Radial Approach in Coronary Chronic Total Occlusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Atadek2017/13
Record Dates: First submitted 2017-08-27; First posted 2017-08-29 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Chronic Coronary Occlusion
Keywords: Femoral approach; Radial approach; Chronic total occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transradial approach (Active Comparator): target vessel revascularization via radial access site is labeled as transradial approach
  Interventions: Other: radial access site
- Transfemoral approach (Active Comparator): target vessel revascularization via femoral access site is labeled as transfemoral approach
  Interventions: Other: femoral access site

INTERVENTIONS:
Other: radial access site — radial route
  Arms: Transradial approach
Other: femoral access site — femoral route
  Arms: Transfemoral approach

SUMMARY:
Pecutaneous coronary intervention (PCI) of chronic total occlusions (CTOs) is most commonly performed using bilateral transfemoral access and 8 French guiding catheters. However, transfemoral approach (TFA) is associated with higher risk of vascular access complications.5 It has been reported that using transradial approach (TRA) reduces vascular complications and may be associated with a better clinical outcome. Transradial access is also used in complex PCI interventions.There is a growing body of evidence regarding the use of this approach also in CTO procedures. In available literature, all studies comparing TRA vs. TFA in CTO consisted of single center and single operator experience. Besides, none of them is randomized. To fill in the gap, we sought to examine the technique and outcomes of transradial vs. transfemoral CTO PCI in a contemporary multicenter randomized study.

DETAILED DESCRIPTION:
All consecutive patients referred for CTO PCI between August 2017 and July 2021 at Acibadem University Kocaeli Acibadem Hospital, Kocaeli; Erciyes University Medical Faculty, Kayseri; Istanbul University Cerrahpasa Medical Faculty, Haseki Cardiology Institute; Istanbul; Memorial Bahcelievler Hospital, Istanbul were screened for enrollment in the study. The exclusion criteria included: (a) any acute coronary syndrome within 3 months; (b) severe heart failure issues; (c)severe renal failure (d) failure to provide written informed consent.The radial access group consisted of patients with single or bi-radial approach. Any femoral artery puncture was considered a femoral case. For example, a crossover from any radial to femoral access was considered a femoral case. Procedures were performed by 4 interventional cardiologists, who are dedicated radial operators, at 4 different centers. The protocol was approved by the institutional review board and all patients provided written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with coronary total occlusion >3 months and indication for intervention

Exclusion Criteria:

* Acute coronary syndrome within 3 months

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
Procedural success | 24 hours
  Technical success without any in-hospital event

SECONDARY OUTCOMES:
Major access site complications | 24 hours
  Major bleeding, vascular complication requiring intervention and hematomas ≥ 10 cm

CONTACTS AND LOCATIONS:
Overall Officials: Sevket Gorgulu, MD, Study Chair — Acibadem University
Locations (4):
- Turkey (Türkiye) (4):
  - Acibadem University, Istanbul
  - Haseki Cradiology Institute, Istanbul
  - Memorial Hospital, Istanbul
  - Erciyes University, Kayseri

REFERENCES:
- [Derived] Gorgulu S, Kalay N, Norgaz T, Kocas C, Goktekin O, Brilakis ES. Femoral or Radial Approach in Treatment of Coronary Chronic Total Occlusion: A Randomized Clinical Trial. JACC Cardiovasc Interv. 2022 Apr 25;15(8):823-830. doi: 10.1016/j.jcin.2022.02.012. PMID 35450683